CLINICAL TRIAL: NCT04500574
Title: Latanoprost Eluting Contact Lens for Treating Glaucoma and Ocular Hypertension
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low recruitment
Sponsor: Massachusetts Eye and Ear Infirmary (Other)
Collaborators: Harvard University (Other)
Responsible Party: Principal Investigator, David Steven Friedman, MD, PhD, MPH, Director Glaucoma Services, Massachusetts Eye and Ear Infirmary
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2020P001916; 2020A000354 (Other Grant/Funding Number: President and Fellows of Harvard College)
Record Dates: First submitted 2020-07-28; First posted 2020-08-05 (Actual); Last update posted 2025-10-15 (Actual); Status verified 2025-10

CONDITIONS: Glaucoma; Ocular Hypertension
Keywords: Latanoprost; Glaucoma; Ocular Hypertension; Drug eluting contact lens
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Latanoprost

STUDY DESIGN:
Intervention Model Description: This is a single-center study to assess the safety and feasibility of delivering latanoprost using the latanoprost contact lens (L-CL) delivery system as a treatment for glaucoma or ocular hypertension. The study has two phases. Phase A is an open-label study with 5 participants; these individuals will wear the L-CL in one eye for one week during which time they will be closely followed with examinations for evaluation of safety. If the L-CL is found to be safe after review of the clinical data by a data and safety monitoring board, phase B will be initiated to assess the safety and effectiveness of delivering latanoprost through the L-CL. This is a double-masked double-dummy study. The L-CL arm will have the drug-eluting latanoprost contact lens (L-CL) and a sham drop, and the latanoprost arm will have a C-CL (no drug) with a nightly 0.005% latanoprost drop.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Latanoprost contact lens (Experimental): The L-CL arm will have the drug-eluting latanoprost contact lens (L-CL) and a sham drop.
  Interventions: Drug: Latanoprost eluting contact lens
- Topical Latanoprost (Placebo Comparator): The placebo arm will have a commercial contact lens with no drug with a nightly 0.005% latanoprost drop.
  Interventions: Drug: Topical Latanoprost

INTERVENTIONS:
Drug: Latanoprost eluting contact lens — The latanoprost-contact lens will be worn in one eye for one week.
  Arms: Latanoprost contact lens
Drug: Topical Latanoprost — A commercial contact lens with no drug will be worn in one eye for one week.
  Arms: Topical Latanoprost

SUMMARY:
In this research study, we will assess the safety, tolerability, comfort, and feasibility of lowering intraocular pressure using a novel Contact Lens Drug Delivery System with latanoprost. Latanoprost is a well-studied medication and has been used to treat glaucoma for decades. Currently, latanoprost is FDA-approved to be administered to patients as eye drops, but using eye drops has challenges (having to remember to take the drop, getting the drop in the eye). This clinical trial is being done to determine the safety, tolerability, and effectiveness of using latanoprost to deliver latanoprost in a new way (through a drug-eluting contact lens).

The study includes two phases. Phase A is intended to assess safety and tolerability and Phase B to assess safety and effectiveness.

DETAILED DESCRIPTION:
In Phase A of this study, five subjects will wear the latanoprost-eluting contact lens (L-CL) for one week. Phase A is designed to assess for safety and tolerability. In Phase B of this research study, we will compare the L-CL to placebo. Patients will be randomized to one of 2 groups. Subjects in Group 1 will receive the contact lens with latanoprost in it (latanoprost contact lens, or "L-CL") and placebo eye drops. Subjects in Group 2 will receive a standard, commercial contact lens (or "C-CL) that contains no latanoprost but will be given latanoprost eye drops. The placebo contact lens (C-CL) is highly similar to the latanoprost-eluting contact lens but contains no latanoprost. The placebo eye drops look just like latanoprost eye drops but contain no latanoprost.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 85 years of age willing and able to give informed consent and in the investigator's judgment able to follow the study protocol
* Ocular hypertension, primary open-angle glaucoma, pigmentary or pseudoexfoliation glaucoma, with mild to moderate glaucoma defined as Mean Deviation on Humphrey Visual Field testing no worse than -10 dB
* Patients on latanoprost in the study eye with an adequate IOP control with latanoprost alone

Exclusion Criteria:

Systemic

* Use of oral carbonic anhydrase inhibitors
* Unstable dose of oral medication during the last 30 days that in the opinion of the Investigator may influence the IOP
* Unstable dose of oral steroid at the time of enrollment
* Use of immunosuppressants, immunomodulators, antimetabolites and/or alkylating agents within six months before screening or anticipated use at any time during the study
* Known allergy or hypersensitivity to the study medication or its components
* Female patients who are pregnant, nursing, or planning a pregnancy, or who are of childbearing potential and not using a reliable means of contraception
* Participation in an investigational drug or device study within the 30 days before screening
* Patient has a condition or is in a situation which, in the Investigator's opinion, may put the patient at significant risk, may confound the study results, or may interfere significantly with the patient's participation in the study
* Any condition (including the inability to read visual acuity charts or language barrier) which precludes a patient's ability to comply with study requirements including completion of the study

Study Eye

* History of complex cataract surgery with vitreous loss
* History of cystoid macular edema or uveitis
* Corneal decompensation or edema
* Corneal thickness <500 or > 600 μm in the study eye by pachymetry
* Prior treatment-related adverse event or allergy to latanoprost
* Evidence of macular edema/intraretinal fluid on screening macula optical coherence tomography (OCT)
* Any ocular condition in the study eye that in the opinion of the investigator would prevent the eye from wearing a contact lens (e.g., ectropion, lid abnormality, or symblepharon)
* Use of beta-blocker, alpha agonist, rho kinase inhibitor, or carbonic anhydrase inhibitor drops within 1 month prior to screening; the use of latanoprost must be stable for at least 4 weeks prior to screening
* Use of latanoprost for < 4 weeks prior to screening
* Use of topical steroids
* Active optic disc or retinal neovascularization in the study eye at screening
* Presence of rubeosis iridis in the study eye at screening
* History of herpetic infection in the study eye or adnexa
* Media opacity in the study eye at screening that precludes clinical and photographic evaluation (including but not limited to preretinal or vitreous hemorrhage, lens opacity)
* Intraocular surgery, including cataract surgery, and/or laser of any type in the study eye within 30 days prior to screening
* History of kerato-refractive surgery
* Any prior filtering surgery, including trabeculectomy, glaucoma drainage device, or Xen implant
* Inability to comfortably wear a commercial contact lens (C-CL) that has the same dimensions as the L-CL during the week-long run-in period

Both Eyes: any active ocular infection (i.e., bacterial, viral, parasitic, or fungal) in either eye at screening

Non-study Eye: Pinhole score < 19 letters (at least 20/400 Snellen equivalent) in the non-study eye at the screening visit

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2024-04-03 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events as assessed by ocular infection, corneal epithelial defects, or cystoid macular edema - Phase A | 6 - 14 weeks
  Safety assessed by the occurrence of the following adverse events: ocular infection, corneal epithelial defects or signs of corneal toxicity that are not contact lens staining patterns, superficial punctate or vortex, cystoid macular edema
Incidence of Treatment-Emergent Adverse Events as assessed by ocular infection, corneal epithelial defects, or cystoid macular edema - Phase B | 6 weeks
  Safety assessed by the occurrence of the following adverse events: ocular infection, corneal epithelial defects or signs of corneal toxicity that are not contact lens staining patterns, superficial punctate or vortex, cystoid macular edema
Efficacy assessed by changes in intraocular pressure - Phase B | 6 weeks
  Effectiveness: % change in intraocular pressure (IOP) from baseline (following washout, i.e., on no medications) in each arm ; Difference in mean intraocular pressure comparing the L-CL arm to the topical latanoprost arm; % change in IOP in each arm compared to baseline IOP on topical latanoprost

SECONDARY OUTCOMES:
Preliminary efficacy - Phase A: % change in IOP from baseline | 6 - 14 weeks
  Assess by comparing % change in IOP from baseline following washout (i.e., on no medications), % change in IOP from topical latanoprost compared to the L-CL
Tolerability and comfort: questionnaire | 6- 14 weeks
  We will assess the tolerability and comfort of the L-CL by using the validated questionnaire Contact Lens Dry Eye Questionnaire-8 (CLDEQ-8). The CLDEQ-8 has as a minimum value a score of 1 and as a maximum value a score of 37. A higher score means a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: David S Friedman, MD, PhD, MPH, Principal Investigator — Massachusetts Eye and Ear
Locations (1):
- Massachusetts Eye and Ear, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available.

REFERENCES:
- [Background] Ciolino JB, Ross AE, Tulsan R, Watts AC, Wang RF, Zurakowski D, Serle JB, Kohane DS. Latanoprost-Eluting Contact Lenses in Glaucomatous Monkeys. Ophthalmology. 2016 Oct;123(10):2085-92. doi: 10.1016/j.ophtha.2016.06.038. Epub 2016 Aug 29. PMID 27586444
- [Background] Ciolino JB, Stefanescu CF, Ross AE, Salvador-Culla B, Cortez P, Ford EM, Wymbs KA, Sprague SL, Mascoop DR, Rudina SS, Trauger SA, Cade F, Kohane DS. In vivo performance of a drug-eluting contact lens to treat glaucoma for a month. Biomaterials. 2014 Jan;35(1):432-9. doi: 10.1016/j.biomaterials.2013.09.032. Epub 2013 Oct 4. PMID 24094935
- [Background] Friedman DS, Wolfs RC, O'Colmain BJ, Klein BE, Taylor HR, West S, Leske MC, Mitchell P, Congdon N, Kempen J; Eye Diseases Prevalence Research Group. Prevalence of open-angle glaucoma among adults in the United States. Arch Ophthalmol. 2004 Apr;122(4):532-8. doi: 10.1001/archopht.122.4.532. PMID 15078671
- [Background] Sleath B, Blalock S, Covert D, Stone JL, Skinner AC, Muir K, Robin AL. The relationship between glaucoma medication adherence, eye drop technique, and visual field defect severity. Ophthalmology. 2011 Dec;118(12):2398-402. doi: 10.1016/j.ophtha.2011.05.013. PMID 21856009